CLINICAL TRIAL: NCT00803959
Title: A Randomized Trial of Urodynamic Testing Before Stress-Incontinence Surgery
Brief Title: Value of Urodynamic Evaluation
Acronym: ValUE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Carelon Research (Other)
Collaborators: University of Alabama at Birmingham (Other); University of California, San Diego (Other); University of Maryland (Other); University of Pittsburgh (Other); University of Texas Southwestern Medical Center (Other); The University of Texas Health Science Center at San Antonio (Other); University of Utah (Other); Beaumont Hospital (Other); Loyola University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ValUE (completed)
Record Dates: First submitted 2008-12-05; First posted 2008-12-08 (Estimated); Results first posted 2013-08-06 (Estimated); Last update posted 2013-08-06 (Estimated); Status verified 2013-07

CONDITIONS: Urinary Incontinence
Keywords: Stress urinary incontinence, Mixed, Urge
MeSH Terms: conditions — Urinary Incontinence; Urinary Incontinence, Stress | interventions — Urodynamics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- No UDS (Active Comparator): Women desiring surgery for diagnosed, uncomplicated predominant stress urinary incontinence (UI) who receive a basic office evaluation only.
  Interventions: Other: Office evaluation
- UDS (Active Comparator): Women desiring surgery for diagnosed, uncomplicated predominant stress urinary incontinence (UI) who receive a basic office evaluation with preoperative urodynamic studies prior to surgery.
  Interventions: Other: Office evaluation; Other: UDS

INTERVENTIONS:
Other: Office evaluation — Office evaluation
Other: UDS — Urodynamics
  Other Names: Urodynamics
  Arms: UDS

SUMMARY:
Although no reliable and specific figures are available for the total expenditure on UDS, UDS is commonly performed for patients with urinary incontinence (UI) regardless of gender and age. UDS is typically performed prior to incontinence surgery. Urodynamic studies are expensive, time-consuming, and uncomfortable diagnostic investigations. The 3rd ICI reported insufficient evidence with which to answer the following key research questions related to UDS: 1) Do physicians alter clinical decision-making based on results of UDS?, and 2) Do alterations in clinical decisions made in response to UDS results improve the clinical outcomes?

ELIGIBILITY:
Inclusion Criteria:

1. Female
2. Predominant SUI as evidenced by all of the following:

   1. Self-reported stress-type UI symptoms, of duration >3 months*
   2. MESA stress symptom score (percent of total possible stress score) greater than MESA urge symptom score (percent of total possible urge score)
3. Observation of leakage by provocative stress test at any volume
4. Eligible for randomization to either treatment group
5. Eligible for SUI surgery
6. Desires non-conservative therapy for SUI
7. PVR <150ml by any method. (May repeat once if initial measure is abnormal)
8. Negative urine dipstick (negative result = trace or less for leukocytes & nitrites) or negative UA or negative culture
9. Available to initiate SUI treatment within 6 weeks of randomization
10. Available for 12-months of follow-up and able to complete study assessments, per clinician judgment.
11. Signed consent form.

    * Patient can be rescreened after respective time interval has been met.

Exclusion Criteria:

1. Age <21 years*
2. Currently undergoing or has had recommended treatment of apical or anterior prolapse
3. No anterior or apical prolapse > +1 on standing straining prolapse exam
4. Pregnant or has not completed child bearing.
5. <12 months post-partum*†
6. Active malignancy of cervix, uterus, fallopian tube(s) or ovary > Stage I, or bladder of any Stage
7. History of pelvic radiation therapy
8. Previous incontinence surgery
9. Current catheter use
10. Neurological disease known to affect bladder storage (e.g. MS, Parkinsonism, CVA)
11. Previous (i.e. repaired) or current urethral diverticulum
12. Prior augmentation cystoplasty or artificial sphincter
13. Implanted nerve stimulators for urinary symptoms or previous botox bladder injections.
14. Any pelvic surgery within the last 3 months*
15. Previous placement of synthetic mesh on a vaginal approach in the anterior compartment
16. Participation in another treatment intervention trial that might influence results of this trial.
17. A urodynamic result reviewed by the investigator in the preceding 12 months or any recollection by the investigator of urodynamic results on that subject.

    * Patient can be rescreened after respective time interval has been met.

      * "Partum" is defined as a delivery or other termination that occurs after 20 weeks gestation.

Min Age: 21 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 630 (Actual)
Dates: Start 2008-11; Primary Completion 2009-12 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ann Gormley, MD, Study Chair — Dartmouth-Hitchcock Medical Center
Locations (10):
- United States (10):
  - University of Alabama, Birmingham, Alabama
  - University of California, San Diego, California
  - Loyola University Medical Center, Maywood, Illinois
  - University of Maryland, Baltimore, Maryland
  - Oakwood Hospital/Cancer Center, Dearborn, Michigan
  - Beaumont Hospital, Royal Oak, Michigan
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - University of Texas Southwestern, Dallas, Texas
  - University of Texas Health Sciences Center, San Antonio, Texas
  - University of Utah, Salt Lake City, Utah

REFERENCES:
- [Background] Nager CW, Brubaker L, Litman HJ, Zyczynski HM, Varner RE, Amundsen C, Sirls LT, Norton PA, Arisco AM, Chai TC, Zimmern P, Barber MD, Dandreo KJ, Menefee SA, Kenton K, Lowder J, Richter HE, Khandwala S, Nygaard I, Kraus SR, Johnson HW, Lemack GE, Mihova M, Albo ME, Mueller E, Sutkin G, Wilson TS, Hsu Y, Rozanski TA, Rickey LM, Rahn D, Tennstedt S, Kusek JW, Gormley EA; Urinary Incontinence Treatment Network. A randomized trial of urodynamic testing before stress-incontinence surgery. N Engl J Med. 2012 May 24;366(21):1987-97. doi: 10.1056/NEJMoa1113595. Epub 2012 May 2. PMID 22551104
- [Result] Nager CW, Brubaker L, Daneshgari F, Litman HJ, Dandreo KJ, Sirls L, Lemack GE, Richter HE, Leng W, Norton P, Kraus SR, Chai TC, Chang D, Amundsen CL, Stoddard AM, Tennstedt SL; Urinary Incontinence Treatment Network. Design of the Value of Urodynamic Evaluation (ValUE) trial: A non-inferiority randomized trial of preoperative urodynamic investigations. Contemp Clin Trials. 2009 Nov;30(6):531-9. doi: 10.1016/j.cct.2009.07.001. Epub 2009 Jul 25. PMID 19635587
- [Derived] Norton PA, Nager CW, Brubaker L, Lemack GE, Sirls LT, Holley R, Chai TC, Kraus SR, Zyczynski H, Smith B, Stoddard A; Urinary Incontinence Treatment Network. The cost of preoperative urodynamics: A secondary analysis of the ValUE trial. Neurourol Urodyn. 2016 Jan;35(1):81-4. doi: 10.1002/nau.22684. Epub 2014 Oct 18. PMID 25327775
- See also: UITN Public Website — http://www.uitn.net

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between November 2008 and June 2010, a total of 630 women underwent randomization (315 in each group) at 11 participating US sites. Of the 53 participating surgeons, 38 were urogynecologists and 15 were urologists; more than 90% were fellowship-trained.
Pre-assignment Details: 4083 women with urinary incontinence were screened for eligibility; of these 2708 did not meet inclusion criteria, 379 declined to participate and 313 were eligible but excluded for administrative reasons. This left 683 who provided written informed consent; 40 were deemed ineligible before randomization and 13 withdrew consent with 630 randomized.
Groups:
- Office Evaluation Only (no UDS): UDS is not conducted during office evaluation visit prior to surgery for women desiring surgery for diagnosed, uncomplicated predominant stress urinary incontinence.
- Urodynamic Testing (UDS Arm): UDS is conducted during office evaluation visit prior to surgery for women desiring surgery for diagnosed, uncomplicated predominant stress urinary incontinence.
Period: Overall Study
Arm/Group | Office Evaluation Only (no UDS) | Urodynamic Testing (UDS Arm)
Started | 315 | 315
ITT Analysis With Primary Outcome Data | 266 | 272
Completed | 259 (Because it is a non-inferiority trial, the PP analysis was the main analysis (n=259).) | 264 (Because it is a non-inferiority trial, the PP analysis was the main analysis (n=264).)
Not Completed | 56 | 51

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Office Evaluation Only (no UDS) | Urodynamic Testing (UDS Arm) | Total
Number analyzed (Participants) | 259 | 264 | 523
Age Continuous [Mean (Standard Deviation); unit: years] | 51.6 (10.0) | 51.9 (10.4) | 51.7 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 259 | 264 | 523
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 259 | 264 | 523

OUTCOME MEASURES:

1. Primary Outcome: Self-reported Urinary Incontinence, Irritative and Obstructive Symptoms: Reduction of 70%+ in the Urogenital Distress Inventory From Baseline to 12 Mos and "Very Much" or "Much" Better on the Patient Global Impression of Improvement Measure at 12 Mos.
Description: Treatment success is defined as a reduction in the Urogenital Distress Inventory score from baseline to 12 months of 70% or more and a Patient Global Impression of Improvement response of "very much better" or "much better" at 12 months.
Time Frame: 12 Months
Population: There were 315 women randomized to each of the arms. In the no UDS arm (and UDS arm), 49 (43) did not have primary outcome data, leaving 266 (272) included in the ITT analysis. Of these, 259 (264) were included in the PP analysis with primary outcome data. The PP analysis was the primary analysis because the outcome was a non-inferiority endpoint.
Measure: Number; unit: percentage of participants
Arm/Group | Office Evaluation Only (no UDS) | Urodynamic Testing (UDS Arm)
Number analyzed (Participants) | 259 | 264
percentage of participants | 77.2 | 76.9
Statistical Analysis 1: Comparison: Office Evaluation Only (no UDS) vs Urodynamic Testing (UDS Arm); The null hypothesis was that the no UDS group was non-inferior to those in the UDS group. Assuming a significance level of 5% and a true success rate in each group of 70% with a noninferiority margin of 11 percentage points, we needed to enroll 270 women/group to have 80% power for determining whether the results in the no UDS group were non inferior to those in the UDS group. Assuming a 10% dropout rate, a sample of 300 women per group was required; Test type: Non-Inferiority or Equivalence — The investigators selected the 11% noninferiority margin on the basis of clinical judgement that it was a reasonable threshold for a trade-off between a decrease in the rate of successful treatment and the potential benefits of eliminating UDS studies from preoperative assessment. To minimize bias toward noninferiority, only women treated per protocol (e.g. who underwent the randomly assigned evaluation) were considered in the primary outcome analysis (ITT analysis considered secondary); Chi-squared; Noninferiority declared if the upper boundary of the two-sided 95% confidence interval for the difference in % success (UDS - no UDS) was < 11%; Difference in success % (UDS - no UDS) = -0.3, 95% CI 2-sided [-7.5 to 6.9] — Point estimates of success percentage are calculated as 200/259= 77.2% for Office Evaluation Only and 203/264 = 76.9% for Urodynamic Testing arm

2. Secondary Outcome: Percentage Meeting or Exceeding 70% Decrease in UDI Score Between Baseline and 12 Months
Description: The Urogenital Distress Inventory is a 20-item patient-reported measure that assesses the presence of urinary incontinence, urgency, frequency, and voiding dysfunction and the extent to which the patient is bothered by these symptoms. Scores range from 0 to 300, with higher scores indicating greater distress. The 70% cutoff value was selected on the basis of the previous experience of the study investigators and receiver-operating- characteristic curve analyses from a previous surgical trial.
Time Frame: Baseline, 12 mos
Population: There were 315 women randomized to each arm. In the UDS arm, 43 did not have primary outcome data leaving 272 in the intention-to-treat group. In the no UDS arm, 49 did not have primary outcome data leaving 266 in the ITT group. ITT analysis was used for all outcomes with the exception of the primary non-inferiority endpoint.
Measure: Number; unit: percentage of participants
Arm/Group | Office Evaluation Only (no UDS) | Urodynamic Testing (UDS Arm)
Number analyzed (Participants) | 266 | 272
percentage of participants | 78.9 | 77.2
Statistical Analysis 1: Comparison: Office Evaluation Only (no UDS) vs Urodynamic Testing (UDS Arm); Null hypothesis is that the two groups will not differ in the percent meeting 70% reduction in Urogenital Distress Inventory score; Test type: Superiority or Other; p = 0.63, Chi-squared — The p-value is not adjusted for multiple comparisons. Alpha level is considered to be 0.05; No adjustments were made; test had 1 degree of freedom

3. Secondary Outcome: Patient Global Impression Index
Description: Patient Global Impression of Improvement is a patient-reported measure of perceived improvement that is obtained by asking study participants, "How is your urinary tract condition now, as compared with how it was before you received treatment for your urinary leakage?" Responses are on a 7-point scale from 1 meaning "very much better" to 7 meaning "very much worse." Values of "very much better" (1) or "much better" (2) were considered to have "perceived improvement" according to this criteria. Values of 3 or greater were not (e.g. "a little better", "no change", "a little worse", "much worse" or "very much worse"). This instrument correlates with the frequency of incontinence episodes, pad tests, and quality of life as it relates to incontinence.
Time Frame: 12 Months
Population: 315 women were randomized to each arm. In the UDS arm, 43 did not have primary outcome data leaving 272 in the intention-to-treat group. In the no UDS arm, 49 did not have primary outcome data leaving 266 in the ITT group. Two were missing PGI-I data in the UDS arm and 4 in the no UDS arm; sample size was 262 in no UDS arm and 270 in the UDS arm.
Measure: Number; unit: percentage of participants
Arm/Group | Office Evaluation Only (no UDS) | Urodynamic Testing (UDS Arm)
Number analyzed (Participants) | 262 | 270
percentage of participants | 90.8 | 91.9
Statistical Analysis 1: Comparison: Office Evaluation Only (no UDS) vs Urodynamic Testing (UDS Arm); Null hypothesis is that there is no difference in the proportion responding "very much better" or "much better" on the Patient Global Impression of Improvement at the 12 month visit; Test type: Superiority or Other; p = 0.68, Chi-squared — P-value not adjusted for multiple comparisons; a priori threshold for statistical significance set at alpha = 0.05; No adjustments made; 1 degree of freedom test

4. Secondary Outcome: Change in Bother as Measured by the UDI
Description: The Urogenital Distress Inventory is a 20-item patient-reported measure that assesses the presence of urinary incontinence, urgency, frequency, and voiding dysfunction and the extent to which the patient is bothered by these symptoms. Scores range from 0 to 300, with higher scores indicating greater distress. Change was calculated as the score at 12 months minus the score at baseline. Higher scores indicate worse function, so the larger the negative value, the greater the improvement.
Time Frame: Baseline, 12 Months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Office Evaluation Only (no UDS) | Urodynamic Testing (UDS Arm)
Number analyzed (Participants) | 266 | 272
units on a scale | -98.4 (51.4) | -100.2 (50.1)
Statistical Analysis 1: Comparison: Office Evaluation Only (no UDS) vs Urodynamic Testing (UDS Arm); Null hypothesis is that the two arms do not differ according to change in UDI score; Test type: Superiority or Other; p = 0.68, t-test, 2 sided — P-value is not adjusted for multiple comparisons; a priori threshold for statistical significance was set at alpha = 0.05; One df t test assumed equal variance; no evidence was found to the contrary

5. Secondary Outcome: Change in Severity as Measured by the ISI
Description: Incontinence Severity Index has scores ranging from 1 to 12 and higher scores indicating greater severity. Change was calculated as the score at 12 months minus the score at baseline. Higher scores indicate worse function, so the larger the negative value, the greater the improvement.
Time Frame: Baseline & 12 Months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Office Evaluation Only (no UDS) | Urodynamic Testing (UDS Arm)
Number analyzed (Participants) | 266 | 272
units on a scale | -5.7 (3.4) | -6.0 (3.3)
Statistical Analysis 1: Comparison: Office Evaluation Only (no UDS) vs Urodynamic Testing (UDS Arm); Null hypothesis is that the 2 arms do not differ according to change in ISI score; Test type: Superiority or Other; p = 0.40, t-test, 2 sided — P-value was not adjusted for multiple comparisons; a priori threshold for statistical significance set at alpha = 0.05; Test was 1 df t-test assuming equal variances; no evidence to the contrary was found

6. Secondary Outcome: Change in MESA Stress Score
Description: The Medical, Epidemiological, and Social Aspects of Aging (MESA) stress score was measured at baseline and the 12 month visit with a possible range from 0 to 100 with higher scores indicating worse function. The outcome measures is change from baseline to 12 mo visit in MESA stress score. Change was calculated as the score at 12 months minus the score at baseline and could range from -100 to 100. Higher raw scores indicate worse function, so the larger the negative change score value, the greater the improvement.
Time Frame: Screen & 12 Months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Office Evaluation Only (no UDS) | Urodynamic Testing (UDS Arm)
Number analyzed (Participants) | 266 | 272
units on a scale | -60.2 (24.7) | -61.5 (22.0)
Statistical Analysis 1: Comparison: Office Evaluation Only (no UDS) vs Urodynamic Testing (UDS Arm); Null hypothesis is that the 2 arms do not differ in change in MESA stress score; Test type: Superiority or Other; p = 0.50, t-test, 2 sided — P-value not adjusted for multiple comparisons; a priori threshold was alpha = 0.05; The t test had 1 df assuming equal variances; no evidence of unequal variances was found

7. Secondary Outcome: Change in MESA Urge Score
Description: The Medical, Epidemiological, and Social Aspects of Aging (MESA) urge score was measured at baseline and the 12 month visit with a possible range from 0 to 100 with higher scores indicating worse function. The outcome measures is change from baseline to 12 mo visit in MESA urge score. Change was calculated as the score at 12 months minus the score at baseline and could range from -100 to 100. Higher raw scores indicate worse function, so the larger the negative change score value, the greater the improvement.
Time Frame: Screen & 12 Months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Office Evaluation Only (no UDS) | Urodynamic Testing (UDS Arm)
Number analyzed (Participants) | 266 | 272
units on a scale | -22.2 (22.4) | -19.7 (21.4)
Statistical Analysis 1: Comparison: Office Evaluation Only (no UDS) vs Urodynamic Testing (UDS Arm); Null hypothesis is that the two arms do not differ according to change in MESA urgency score; Test type: Superiority or Other; p = 0.19, t-test, 2 sided — P-value not adjusted for multiple comparisons and a priori threshold for statistical significance set at alpha = 0.05; The t test had 1 df and assumed equal variances; no evidence of different variances was found

8. Secondary Outcome: Change in Quality of Life as Measured by the IIQ
Description: Incontinence Impact Questionnaire has scores ranging from 0 to 400 and higher scores indicating a more negative effect on quality of life. Change was calculated as the score at 12 months minus the score at baseline and scores could range from -400 to 400. Higher scores indicate worse function, so the larger the negative value, the greater the improvement.
Time Frame: Baseline, 12 Months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Office Evaluation Only (no UDS) | Urodynamic Testing (UDS Arm)
Number analyzed (Participants) | 266 | 272
units on a scale | -37.3 (23.7) | -35.9 (23.2)
Statistical Analysis 1: Comparison: Office Evaluation Only (no UDS) vs Urodynamic Testing (UDS Arm); Null hypothesis is that the 2 arms do not differ according to mean change in IIQ score; Test type: Superiority or Other; p = 0.49, t-test, 2 sided — P-value not adjusted for multiple comparisons and a priori threshold for statistical significance set at alpha = 0.05; T test had 1 df and assumed equal variance; no evidence of different variances was found

9. Secondary Outcome: Change in Quality of Life as Measured by the SF-12
Description: The Medical Outcomes Study 12-Item Short Form Health Survey has scores ranging from 0 to 200 and higher scores indicating better health. Change was calculated as the score at 12 months minus the score at baseline and could range from -200 to 200. The larger the positive value, the greater the improvement.
Time Frame: Baseline, 12 Months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Office Evaluation Only (no UDS) | Urodynamic Testing (UDS Arm)
Number analyzed (Participants) | 266 | 272
units on a scale | 7.3 (12.0) | 5.0 (10.8)
Statistical Analysis 1: Comparison: Office Evaluation Only (no UDS) vs Urodynamic Testing (UDS Arm); Null hypothesis is that the 2 arms do not differ according to mean change in SF-12 scores; Test type: Superiority or Other; p = 0.02, t-test, 2 sided — P-value not adjusted for multiple comparisons and a priori threshold for statistical significance set at alpha = 0.05; T test had 1 df assuming equal variances; no evidence of unequal variances was found

10. Secondary Outcome: Change in Severity as Measured by the PGI-S
Description: The Patient Global Impression of Severity has scores ranging from 1 [normal] to 4 [severe]. Change was calculated as the score at 12 months minus the score at baseline and could range from -3 to 3. Higher scores indicate worse function, so the larger the negative value, the greater the improvement.
Time Frame: Baseline & 12 Months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Office Evaluation Only (no UDS) | Urodynamic Testing (UDS Arm)
Number analyzed (Participants) | 266 | 272
units on a scale | -1.8 (0.9) | -1.8 (0.9)
Statistical Analysis 1: Comparison: Office Evaluation Only (no UDS) vs Urodynamic Testing (UDS Arm); Null hypothesis is that the 2 arms do not differ according to mean change in PGI-S score; Test type: Superiority or Other; p = 0.51, t-test, 2 sided; The t test had 1 df and assumed equal variance; no evidence of different variances was found

11. Secondary Outcome: Moderate or Severe Severity as Measured by the PGI-S
Description: The Patient Global Impression of Severity (PGI-S) has scores ranging from 1 [normal] to 4 [severe]. This measure is the percentage of participants responding to the PGI-S with a "3" corresponding to the "moderate" category or a "4" corresponding to the "severe" category at the 12 month visit.
Time Frame: 12 Months
Population: There were 315 women randomized to each arm. In the UDS arm, 43 did not have primary outcome data leaving 272 in the intention-to-treat group. In the no UDS arm, 49 did not have primary outcome data leaving 266 in the ITT group. One woman was missing PGI-S data in the UDS arm and was excluded leaving n=271 in the UDS arm.
Measure: Number; unit: percentage of participants
Arm/Group | Office Evaluation Only (no UDS) | Urodynamic Testing (UDS Arm)
Number analyzed (Participants) | 266 | 271
percentage of participants | 5.6 | 7.0
Statistical Analysis 1: Comparison: Office Evaluation Only (no UDS) vs Urodynamic Testing (UDS Arm); Null hypothesis is that the 2 arms do not differ in the proportion of women who score moderate or severe on the PGI-S at 12 months; Test type: Superiority or Other; p = 0.51, Chi-squared; Chi-squared test had 1 df and no adjustments

12. Secondary Outcome: Patient Satisfaction With Treatment Outcome
Description: A summary score for patient satisfaction was based on responses to questions developed for this study with scores ranging from 0 to 100 and higher scores indicating better satisfaction.
Time Frame: 12 Months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Office Evaluation Only (no UDS) | Urodynamic Testing (UDS Arm)
Number analyzed (Participants) | 266 | 272
units on a scale | 82.2 (28.6) | 79.5 (30.4)
Statistical Analysis 1: Comparison: Office Evaluation Only (no UDS) vs Urodynamic Testing (UDS Arm); Null hypothesis is that the 2 arms do not differ according to mean overall patient satisfaction score at 12 months; Test type: Superiority or Other; p = 0.28, t-test, 2 sided — P-value was not adjusted for multiple comparisons and the a priori threshold for statistical significance was alpha = 0.05; T test had 1 df and assumed equal variances; no evidence of unequal variances was found

13. Secondary Outcome: Stress Test at 12 Mos
Description: A provocative stress test at a bladder volume of 300 ml was performed for direct observation of urine leakage. Observed urine loss from the urethra coincidental with the Valsalva maneuver or cough was considered a positive test. The stress test was not performed by the study surgeon but rather by an outcome assessor who was unaware of the study assignments.
Time Frame: Screen and 12 months
Population: There were 315 women randomized to each arm. In the UDS arm, 43 did not have primary outcome data leaving 272 in the intention-to-treat group. In the no UDS arm, 49 did not have primary outcome data leaving 266 in the ITT group. Of these, only 225 in the UDS arm and 222 in the no UDS had stress test data at 12 months.
Measure: Number; unit: percentage of participants
Arm/Group | Office Evaluation Only (no UDS) | Urodynamic Testing (UDS Arm)
Number analyzed (Participants) | 222 | 225
percentage of participants | 11.7 | 16.0
Statistical Analysis 1: Comparison: Office Evaluation Only (no UDS) vs Urodynamic Testing (UDS Arm); Null hypothesis is that the proportion having a positive provocative stress test at 12 months was the same in both treatment arms; Test type: Superiority or Other; p = 0.19, Chi-squared — P-values was not adjusted for multiple comparisons and the a priori threshold for statistical significance was set at alpha = 0.05; Chi-squared test had 1 df and no adjustments

ADVERSE EVENTS:
Arm/Group | Office Evaluation Only (no UDS) | Urodynamic Testing (UDS Arm)
Serious Adverse Events (participants affected / at risk) | 30/315 | 21/315
Other Adverse Events (participants affected / at risk) | 39/315 | 49/315
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Office Evaluation Only (no UDS) (N=315) | Urodynamic Testing (UDS Arm) (N=315)
Bladder Perforation (Surgical and medical procedures) | 18 (18) | 12 (12)
Intraoperative Bleeding (Surgical and medical procedures) | 0 (0) | 1 (1)
Mesh complication: erosion (Surgical and medical procedures) | 1 (1) | 0 (0)
Mesh complication: exposure (Surgical and medical procedures) | 3 (3) | 2 (2)
Recurrent UTI (Infections and infestations) | 3 (3) | 1 (1) — Recurrent UTI is defined as presumed UTI with treatment, 3 or more in one year after 6 weeks post surgery with no time limit for reporting.
Granulation Tissue (Surgical and medical procedures) | 0 (0) | 1 (1)
Voiding dysfunction (Renal and urinary disorders) | 5 (5) | 3 (3)
Other: Fascial Wound Dehiscence (Surgical and medical procedures) | 1 (1) | 0 (0)
Other: Vaginal Perforation with sling (Surgical and medical procedures) | 0 (0) | 1 (1)
Other: episode of postoperative bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Office Evaluation Only (no UDS) (N=315) | Urodynamic Testing (UDS Arm) (N=315)
Anesthetic Complication (Surgical and medical procedures) | 0 (0) | 3 (3)
Intraoperative Bleeding (Surgical and medical procedures) | 1 (1) | 2 (2)
Postoperative bleeding (Surgical and medical procedures) | 1 (1) | 2 (2)
Mesh complication: erosion (Surgical and medical procedures) | 1 (1) | 1 (1)
Mesh complication: exposure (Surgical and medical procedures) | 4 (5) | 2 (2)
Surgical site infection: superficial incisional (Surgical and medical procedures) | 1 (1) | 1 (1)
Surgical site infection: deep incisional (Surgical and medical procedures) | 1 (1) | 0 (0)
Surgical site infection: organ/space (Surgical and medical procedures) | 0 (0) | 1 (1)
Culture proven UTI (Infections and infestations) | 13 (14) | 15 (15)
Empiric UTI (Infections and infestations) | 12 (12) | 11 (11)
Recurrent UTI (Infections and infestations) | 0 (0) | 3 (3)
Granulation tissue (Surgical and medical procedures) | 2 (2) | 2 (2)
Voiding dysfunction (Renal and urinary disorders) | 1 (1) | 3 (3)
Other (General disorders) | 9 (9) | 12 (12)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No